CLINICAL TRIAL: NCT06249867
Title: A Randomized, Double-blind, Single Center, Phase 2 Study to Assess the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of 15 mg of Darifenacin Daily in Patients With Amyotrophic Lateral Sclerosis
Brief Title: A Study to Assess the Safety, Tolerability, and Pharmacology of Darifenacin in Patients With ALS
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Oliver Blanchard (Other)
Collaborators: Université de Montréal (Other)
Responsible Party: Sponsor-Investigator, Oliver Blanchard, Assistant Professor, McGill University
Organization: McGill University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ALS-DARI-1
Record Dates: First submitted 2024-01-22; First posted 2024-02-08 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2024-11

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: Amyotrophic lateral sclerosis; Darifenacin; Neuromuscular junction
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — darifenacin

STUDY DESIGN:
Intervention Model Description: Participants are assigned to either a treatment (darifenacin) or placebo group in parallel for the duration of the study. Treatment will include a two-week titration period with a 7.5 mg dose of darifenacin, which will be increased to 15 mg dose for the following 22 weeks. Dosing regimen of the placebo group will be administered to match the treatment dosing regimen.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Darifenacin Treatment (Experimental): Patients in the Treatment arm will receive a daily dose of 1 or 2 darifenacin extended-release tablets.
  Interventions: Drug: Darifenacin 7.5 MG Extended Release Oral Tablet
- Placebo (Placebo Comparator): Patients in the Placebo arm will receive a daily dose of 1 or 2 placebo tablets.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Darifenacin 7.5 MG Extended Release Oral Tablet — During the first two weeks (titration period), patients in the treatment arm will receive a daily dose of 7.5 mg darifenacin extended-release tablet. After the titration period, the dose will be increased to 15 mg once daily, which consists of two 7.5 mg tablets together for a period of 22 weeks.
  Other Names: Darifenacin
  Arms: Darifenacin Treatment
Drug: Placebo — During the first two weeks (titration period), patients in the placebo arm will receive a daily dose of 1 placebo tablet. After the titration period, the dose will be increased to two placebo tablets taken together, for a period of 22 weeks.
  Arms: Placebo

SUMMARY:
Amyotrophic lateral sclerosis (ALS) is a progressive neurological disorder characterized by selective death of upper and lower motor neurons, which leads to severe disability and fatal outcomes. One of the major hallmarks of ALS is the denervation of neuromuscular junctions (NMJs), which is one of the earliest events seen in ALS patients and mouse models of ALS. Under healthy conditions, glial cells called Perisynaptic Schwann Cells (PSCs) have a key role in regulating the stability and maintenance of NMJs, but they only participate in NMJ repair once denervation occurs. Denervation and the subsequent decline in synaptic activity triggers a loss of muscarinic acetylcholine receptors (mAChRs) in the PSC, and the resulting decrease in mAChR-mediated gene expression drives the "repair mode" of the PSC. In assessing the NMJ under conditions of ALS, a scarcity of process extensions in PSCs was observed for months prior to disease onset in the superoxide dismutase 1 (SOD1) mouse model of ALS, indicating inadequate glial repair. Collectively, these preclinical findings support the hypothesis that dampening glial mAChRs will restore the anticipated "repair" response of PSCs in the NMJ. Hence, the use of a selective M3 muscarinic receptor antagonist, Darifenacin, as a disease-modifying therapeutic in familial and sporadic ALS could improve NMJ function, resulting in a beneficial impact on the autonomy and quality of life of ALS patients.

The purpose of the current Phase 2 trial is therefore to test the safety, tolerability, and pharmacology of Darifenacin in patients with ALS. Specifically, 30 eligible subjects between 18 and 85 years of age will take 7.5 mg of darifenacin or placebo daily (by mouth) for two weeks followed by an increased dose of 15 mg for the next 22 weeks. The trial will evaluate the effects of this medication on several outcome measures including patient safety, physical and neurological function, muscle strength, depression levels, and NMJ innervation of patients with ALS. Detailed clinical assessments will be conducted at regular intervals throughout the study in order to achieve these objectives.

DETAILED DESCRIPTION:
ALS is a rapidly progressive neurodegenerative disorder caused by the selective death of motor neurons within the brain, brainstem, and spinal cord, leading to paralysis and death within 2-5 years after diagnosis. A limited number of disease-modifying treatments are available for patients with ALS, namely Riluzole (Rilutek), Edaravone (Radicava), and AMX0035 (Relyvrio in the USA and Albrioza in Canada), and novel therapeutic approaches are being investigated to tackle several aspects of ALS pathological features.

One of the major hallmarks of ALS is the denervation of neuromuscular junctions (NMJs), which is one of the earliest events seen in ALS patients and murine models that recapitulate ALS-like aspects of the disease due to ALS-causing mutations in the SOD1, TDP-43, and FUS genes. It has been shown that an extensive and extended period of NMJ denervation-reinnervation cycles occurs months prior to disease onset in SOD1 ALS mice. To be specific, scarce Perisynaptic Schwann Cell (PSC) process extensions were observed, which indicates inadequate glial repair. Therefore, while PSCs are responsive to NMJ alterations in ALS, their response does not support NMJ repair. PSCs have a key role in regulating the stability and maintenance of NMJs. They actively participate in NMJ repair once denervation and loss of muscarinic acetylcholine receptors (mAChRs) occur. Additionally, regulation of PSC gene expression, governed by mAChR activation, drives the dynamic adaptation of the PSC in a synaptic activity-dependent manner. PSCs will switch to a repair mode when mAChR activation is reduced, such as following a sciatic nerve crush injury and during synapse formation.

Collectively, these preclinical findings support the hypothesis that dampening glial mAChRs will restore the anticipated "repair" response of PSCs in the NMJ. Hence, the use of a selective M3 muscarinic receptor antagonist, Darifenacin, as a disease-modifying therapeutic in familial and sporadic ALS could improve NMJ function, resulting in a beneficial impact on the autonomy and quality of life of ALS patients. The purpose of the current Phase 2 trial is therefore to test the safety, tolerability, and pharmacology of Darifenacin in patients with ALS.

APO-DARIFENACIN (Darifenacin Extended Release Tablets), darifenacin as darifenacin hydrobromide, is a known active substance with the chemical name: (S)-2-{1-[2-(2,3-Dihydrobenzofuran-5-yl)ethyl]-3-pyrrolidnyl}-2,2-diphenylacetamide hydrobromide. For the purposes of this trial, darifenacin has been formulated by Apotex Inc. as an extended release tablet. Darifenacin will be produced and formulated into 7.5 mg coated tablets (extended-release) and a placebo film-coated tablet will be manufactured without the active substance.

Patient enrollment for this trial will consist of 30 eligible ALS patients between 18 and 85 years of age. During the first two weeks (titration period), patients will receive a daily dose of either a placebo or a 7.5 mg darifenacin extended-release tablet. After the titration period, the dose will be increased to 15 mg once daily, which consists of two 7.5 mg tablets together. Depending on the patient's response to the medication, they may be asked to temporarily or permanently stop taking the drug or reduce their dose from 15 mg to 7.5 mg for safety reasons. This treatment period has been selected as a standard for phase 2 trials to study the endpoints and observe significant differences in the outcome measures.

The trial will evaluate the effects of this medication and dosing regimen on several outcome measures including patient safety, physical and neurological function, muscle strength, depression levels, and NMJ innervation of patients with ALS. Detailed clinical assessments will be conducted at regular intervals throughout the study in order to achieve these objectives.

ELIGIBILITY:
Inclusion Criteria:

1. Able to comprehend and willing to sign an Informed Consent Form (ICF).
2. Male or female, ≥ 18 years old and ≤85 years old, at the time of signing the ICF.
3. Confirmed diagnosis of familial or sporadic ALS, defined as meeting the probable, laboratory-supported probable, or definite criteria for a diagnosis of ALS according to the World Federation of Neurology Modified El Escorial criteria (1).
4. ALS duration of less than 36 months from the symptom onset.
5. FVC of ≥ 50 %.
6. Able to swallow tablets without crushing.
7. A female patient is eligible to participate if she is not breastfeeding, has negative pregnancy test at screening, has no intention of becoming pregnant during the course of the study, and agrees to use appropriate contraceptive drugs or devices (as defined in section 3.4 of the study protocol) for the duration of the study.
8. If male and has a partner who may become pregnant, agrees to ensure that he and/or his partner use a reliable form of birth control (as defined in section 3.4 of the study protocol) for the duration of the study and refrain from donating sperm during this period.
9. Participants receiving standard care for ALS prior to entering the trial (i.e. Riluzole, Edaravone, and Albrioza), must be on a stable dosing regimen prior to the randomization and agree to remain on this dosage during the study period:

   * In the case of taking Riluzole, the patient must have been on a stable dose at least 30 days prior to start date.
   * In the case of taking Edaravone, the patient must have been on a stable dose at least 30 days prior to start date.
   * In the case of receiving Albrioza, the patient must have been on a stable dose at least 30 days prior to start date.
10. For participants who consent to the optional biopsy:

    * Participants with normal platelet or coagulation test values.
    * Participants who are receiving anticoagulant medications will need to abstain from using anticoagulants for a specific number of days before and after the biopsy, as decided by the study doctor on a case-by-case basis.

Exclusion Criteria:

1. Patients with, or at risk for, the following conditions:

   * Untreated or uncontrolled narrow-angle glaucoma;
   * Gastric retention
   * Urinary retention
   * Liver disease
2. Patients with a known history of severe allergic or anaphylactic reactions to antimuscarinic medications
3. If diagnosed with another neurodegenerative disease (e.g. Multiple Sclerosis, Parkinson, Myasthenia Gravis, and Alzheimer's disease).
4. Subjects with severe hepatic impairment or abnormal liver enzymes, as defined as Child-Pugh B and C scores.
5. Subject has a history of, or positive test result at Screening, for hepatitis C virus antibody.
6. Subjects with acute or prolonged hepatitis B & C.
7. Any medical condition that might interfere with the patient's participation in the trial, poses any added risk for the patient, or confounds the assessment of the patient according to the Investigator's judgement.
8. Subjects with any uncontrolled (unresolved) medical condition other than ALS, as determined by the Investigator.
9. Subjects who are currently enrolled in another clinical trial and receiving an Investigational Product (IP) (including but not limited to stem cell therapy or gene therapy).
10. Treatment with an investigational drug within 1 month or within a time period equal to 5 half-lives (if known) whichever is longer, of starting study treatment.
11. Patients with prior darifenacin treatment.
12. History of drug and/or alcohol abuse (according to Diagnostic and Statistical Manual of Mental Disorders) prior to the screening as determined by the Investigator.
13. If female, subjects who are pregnant, breastfeeding, or intending to conceive during the course of the study.
14. Subjects with an abnormal electrocardiogram (ECG) at screening (any abnormality that the PI believes that entering the study place the participant at risk).
15. Subjects who are receiving strong CYP3A4 inducers such as carbamazepine (anticonvulsant), phenytoin (anticonvulsant), rifampin (antibiotic), and modafinil (wakefulness-promoting agent).
16. Subjects who are receiving potent CYP3A4 inhibitors such as clarithromycin (macrolide antibiotic), ketoconazole and itraconazole (antifungal medications), nefazadone (antidepressant), nelfinavir and ritonavir (protease inhibitors).
17. Subjects who are receiving or received within 30 days prior to the starting of the trial CYP2D6 substrates with a narrow therapeutic window such as include flecainide (Class IC anti-arrhythmic), thioridazine (antipsychotic) and tricyclic antidepressants.
18. Subjects who are receiving or received botulinum injections in the past 6 months.
19. Subjects who are receiving or received within 30 days prior to the starting of the trial antimuscarinic medications for the treatment of overactive bladder such as fesoterodine, oxybutynin, solifenacin, tolterodine, and trospium.
20. Only for patients that consented to the Optional Needle Muscle Biopsy procedures.
21. Subject is taking an anticoagulant (with the exception of aspirin at the investigator's discretion) or is at risk of increased or uncontrolled muscle biopsy-related bleeding.
22. Subjects with bleeding risk factors which include, but are not limited to, anatomical factors at or near the muscle biopsy site (e.g., vascular abnormalities, neoplasms, or other abnormalities) or abnormal platelet or coagulation test values at visit 1.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-11-08 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability of oral doses of 15 mg darifenacin | 24 weeks
  The incidence of adverse events and any abnormal clinical assessments will be monitored.

SECONDARY OUTCOMES:
Pharmacokinetics of oral doses of darifenacin | 4 weeks
  The pharmacokinetic profile of darifenacin in ALS patients will be visualized at Day 1, 14, and 28.
Electrical Impedance Myography (EIM) | 24 weeks
  EIM is a non-invasive technique that measures the electrical impedance characteristics of specific muscles or muscle groups as a readout of muscle health.
Amyotrophic Lateral Sclerosis Functional Rating Scale-Revised (ALSFRS-R) score | 24 weeks
  The ALSFRS-R will be used to measure activities of daily living (ADL) and global function across four domains (respiratory, bulbar function, gross motor skills, and fine motor skills) and consists of 12 questions, each scored from 0 to 4, for a total possible score of 48, with higher scores representing better function.
Forced Vital Capacity (FVC) | 24 weeks
  The FVC test examines lung capacity and overall respiratory function.
King's College (KINGS) stage | 24 weeks
  The KINGS staging system for ALS will be used to assess the course of the disease and is based on the number of involved regions (where the three possible regions are bulbar, upper limb or lower limb) for the first three stages and the need for gastrostomy and non-invasive ventilation for the subsequent stages. The possible stages in the KINGS staging system are as follows: Stage 1: First Region Involved; Stage 2: Second Region Involved; Stage 3: Third Region Involved; Stage 4a: Nutritional Failure (need for gastrostomy); Stage 4b: Respiratory Failure (need for non-invasive ventilation); and Stage 5: Death.
Hand-Held Dynamometry (HHD) | 24 weeks
  HHD will be used to examine muscle strength in various muscles of the arms and legs.
ALS Assessment Questionnaire (ALSAQ5) | 24 weeks
  The ALSAQ-5 is one of the most widely validated measures of health status for use with patients diagnosed with ALS. This questionnaire evaluates 5 subdimensions: mobility, ADL, eating and drinking, communication, and emotional functioning.

OTHER OUTCOMES:
Depression and depressive symptoms | 24 weeks
  The self-administered Patient Health Questionnaire (PHQ-9) will be used to assess depressive symptoms.
Physical function and daily activities | 24 weeks
  The self-administered the Rasch-Built Overall Amyotrophic Lateral Sclerosis Disability Scale (ROADS) questionnaire will assess levels of overall disability in patients.
Neuromuscular junction innervation | 24 weeks
  Neuromuscular junctions (NMJs) will be functionally and visually examined to monitor the effect of darifenacin.
Pharmacodynamics of oral doses of 15 mg darifenacin | 24 weeks
  Blood-based biomarkers will be examined on Day 1, 14, 28, and 168 to determine the pharmacodynamic profile of darifenacin in ALS patients.

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Blanchard, MD, Principal Investigator — McGill University - Montreal Neurological Institute
Locations (2):
- Canada (2):
  - Ottawa Hospital Research Institute, Ottawa, Ontario
  - Montreal Neurological Institute, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No